CLINICAL TRIAL: NCT04888611
Title: Neoadjuvant PD-1 Antibody Alone or Combined With Autologous Glioblastoma Stem-like Cell Antigens-primed DC Vaccines (GSC-DCV) for Patients With Recurrent Glioblastoma：A Phase II, Randomized Controlled, Double Blind Clinical Trial.
Brief Title: Neoadjuvant PD-1 Antibody Alone or Combined With DC Vaccines for Recurrent Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); Shanghai Sunstem Biotechnology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Yu Yao, MD, MD, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2021-547
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Glioblastoma
Keywords: Glioblastoma; PD-1 antibody; DC vaccine; Immunotherapy
MeSH Terms: conditions — Glioblastoma | interventions — camrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant PD-1 inhibitor plus DC vaccine (Experimental): Patients will receive neoadjuvant Camrelizumab (PD-1 antibody), followed by surgical resection, DC vaccines and further PD-1 inhibitor treatment until toxicity or progression.
  Interventions: Biological: Camrelizumab plus GSC-DCV
- Neoadjuvant PD-1 inhibitor plus Placebo (Active Comparator): Patients will receive neoadjuvant Camrelizumab (PD-1 antibody), followed by surgical resection, placebo and further PD-1 inhibitor treatment until toxicity or progression.
  Interventions: Biological: Camrelizumab plus Placebo

INTERVENTIONS:
Biological: Camrelizumab plus GSC-DCV — Prior to scheduled surgery, patients need to receive Camrelizumab IV (3mg/kg, up to 200mg). After surgery, patients receive Camrelizumab IV (3mg/kg, up to 200mg) and GSC-DCV IH every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Arms: Neoadjuvant PD-1 inhibitor plus DC vaccine
Biological: Camrelizumab plus Placebo — Prior to scheduled surgery, patients need to receive Camrelizumab IV (3mg/kg, up to 200mg). After surgery, patients receive Camrelizumab IV (3mg/kg, up to 200mg) and Placebo IH every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Arms: Neoadjuvant PD-1 inhibitor plus Placebo

SUMMARY:
Glioblastoma multiforme (GBM) are the most prevalent malignant tumor in central nervous system. At recurrence, no clear standard-of-care therapy is agreed for recurrent GBM (rGBM) and median overall survival is estimated to rarely exceed 6-9 months with effective therapies. Neoadjuvant therapy with anti-PD-1 monoclonal antibodies were confirmed to be helpful to extend survival in rGBM. Vaccine, dendritic cells (DCs) pulsed with glioblastoma stem-like cell (GSC) antigens (GSC-DCV), could extend survival for GBM patients in our previous clinical study (PMID: 30159779). The purpose of this study is to evaluate the safety and efficiency of using the neoadjuvant therapy with PD-1 antibody (Carilizumab) plus DC vaccine (GSC-DCV) in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
This is a phase II randomized controlled clinical study. The purpose of this research is to study the safety and efficacy of Camrelizumab alone or combined with GSC-DCV vaccines in treating patients with recurrent glioblastomas. The participants will be randomly assigned into two group. Patients in group A will receive neoadjuvant Camrelizumab (PD-1 antibody), followed by surgical resection, DC vaccines and further PD-1 inhibitor treatment until toxicity or progression. Patients in group B will receive neoadjuvant Camrelizumab (PD-1 antibody), followed by surgical resection, placebo and further PD-1 inhibitor treatment until toxicity or progression. Furthermore, to evaluate the associations between exploratory biomarkers, clinical outcomes, and adverse events based on the next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 70 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
3. Estimated life expectancy > 3 months.
4. Previous first-line therapy with radiotherapy and chemotherapy, first or second relapse with unequivocal evidence of tumor progression.
5. Pathological diagnosis or molecular diagnosis for lesion this time was confirmed to be recurrent brain glioma (WHO grade 4).
6. Patients with subtotal resection or above of the tumor confirmed with contrast MR within 72 hours after surgery.
7. No high-dose systemic corticosteroids (defined as >10 mg day-1 of prednisone or bio-equivalent for at least seven consecutive days before administration).
8. No antibiotics for at least three consecutive days before administration.
9. Adequate organ function defined by:

   Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥ 1.0×10^9/L, platelets ≥100×10^9/L; hemoglobin ≥ 8 g/dL. Hepatic: bilirubin 2×upper limit of normal (ULN), aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5×upper limit of normal (ULN). Renal: Normal serum Creatinine for age (below) or creatinine clearance >60 ml/min/1.73 m2. Electrocardiogram: normal.
10. Written informed consent.
11. Patient should have good follow-up compliance.

Exclusion Criteria:

1. Pregnant or breast-feeding patients.
2. Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with history of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, ongoing pregnancy, transplant immuno-suppression), or medication of cortisol.
4. Patients with any conditions that could potentially alter immune function (e.g., AIDS, multiple sclerosis, diabetes, renal failure).
5. Any previous investigational medication within 30 days before first administration of Camrelizumab.
6. History of allergy to study drug components or of severe hypersensitivity reactions to any monoclonal antibodies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 24 months
  Time from enrollment to the dates of death from any cause or last follow up reported
Progression-free survival (PFS) | 12 months
  Time from enrollment to the dates of disease progression, death from any cause or last tumor assessment reported between date of first patient enrollment

SECONDARY OUTCOMES:
Number of treatment-related adverse events | 12 months
  Toxicity assessed by Common Terminology Criteria for Adverse Events
Treatment Responses Rate | 6 months
  Response rate assessed by immunotherapy Response Assessment for Neuro-Oncology (iRANO) criteria

OTHER OUTCOMES:
Exploratory biomarkers | 24 months
  To investigate the association between biomarkers and clinical outcomes using diverse biospecimen based on the next generation sequencing, including ctDNA, TIL (tumor infiltrating lymphocyte) density and TCR (T cell receptor) Clonality, gene expression signature, genomic mutation, microbial bacteria and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China